CLINICAL TRIAL: NCT03267069
Title: Evaluating Alcohol Use in Alcoholic Liver Disease
Status: Recruiting | Type: Observational
Sponsor: Nicole T Shen (Other)
Responsible Party: Sponsor-Investigator, Nicole T Shen, Gastroenterology and Hepatology Fellow Physician, New York Presbyterian Hospital
Organization: New York Presbyterian Hospital (Other)
Other Study IDs: 1601016922
Record Dates: First submitted 2017-08-21; First posted 2017-08-30 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Alcoholic Liver Disease
MeSH Terms: conditions — Liver Diseases, Alcoholic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- alcohol liver disease: Patients with alcohol liver disease consenting to participate in the study will be administered an initial survey at inclusion and then follow-up surveys at 3, 6, 9, 12, 15, and 18 month intervals and then 2, 5, and 10 years. There is no intervention cohort, all enrolled will complete the same surveys. Recidivism will be measured by responses to survey questions, clinical interviews documented in the chart, and urine ethnyl glucuronide or blood ethanol testing.
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — surveys will be administered at inclusion and follow-ups

SUMMARY:
This prospective, analytic observational study will investigate alcohol recidivism in patients with alcoholic liver disease. All adult subjects presenting with alcoholic liver disease are considered for inclusion. Subjects able to give consent are included.

DETAILED DESCRIPTION:
This is a longitudinal observational study. Subjects with a diagnosis of alcoholic liver disease (acute alcoholic hepatitis or alcoholic cirrhosis) who present to Weill Cornell Medical Center or Columbia University Medical Center New York Presbyterian Hospital or the Gastroenterology and Hepatology Clinic will be invited to join this study, which entails a survey at baseline and follow-up at 3, 6, 9, 12, 15, and 18 months and then at 2, 5, and 10 years. Follow-up will consist of a chart review, a phone or in person interview, and most recent clinic visit interview for alcohol recidivism. The clinical providers will be blinded to the survey results.

ELIGIBILITY:
Inclusion Criteria:

* alcoholic liver disease able to consent

Exclusion Criteria:

* without alcoholic liver disease unable to consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects with alcoholic liver disease
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2016-11-27 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
alcohol recidivism assessed by questionnaire | 6 months
  Follow-up questionnaires will be administered at 6 months assessing for alcohol use
alcohol recidivism assessed by clinical interview | 6 months
  Follow-up interviews will be conducted at 6 months assessing for alcohol use
alcohol recidivism assessed by urine ethyl glucuronide | 6 months
  Follow-up urine testing may be conducted at 6 months assessing for alcohol use
alcohol recidivism assessed by blood | 6 months
  Follow-up blood testing may be conducted at 6 months assessing for alcohol use

SECONDARY OUTCOMES:
alcohol recidivism assessed by questionnaire | after 6 months
  Follow-up questionnaires will be administered after 6 months assessing for alcohol use
alcohol recidivism assessed by clinical interview | after 6 months
  Follow-up clinical interviews will be conducted after 6 months assessing for alcohol use
alcohol recidivism assessed by urine ethyl glucuronide | after 6 months
  Follow-up urine testing may be conducted after 6 months assessing for alcohol use
alcohol recidivism assessed by blood | after 6 months
  Follow-up blood testing may be conducted after 6 months assessing for alcohol use

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Brown, MD, MPH, Principal Investigator — New York Presbyterian Hospital - Weill Cornell Medicine and Columbia University Medical Center
Locations (1):
- New York Presbyterian Hospital - Weill Cornell Medicine and Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fahoum K, Shen NT, Basu E, Lee J, Kaplan A, Salajegheh A, Rosenblatt R, Jesudian A, Lucero C, Fortune B, Safford M, Brown RS Jr. Prognostic Factors in Alcohol-associated Liver Disease Patients Presenting With First Evidence of Ascites. J Clin Gastroenterol. 2024 Feb 1;58(2):200-206. doi: 10.1097/MCG.0000000000001836. PMID 37126326